CLINICAL TRIAL: NCT00221273
Title: Randomized Clinical Trial to Assess the Clinical Effectiveness of a Measured Objective Tensioning in Hamstring ACL Reconstruction
Brief Title: Use of Graft Tensioner Device in ACL (Knee) Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H05-70302
Record Dates: First submitted 2005-09-18; First posted 2005-09-22 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Torn Anterior Cruciate Ligament (Knee)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ACL surgery

SUMMARY:
Compares tension of an ACL graft when using a commercial device vs. the tension of the graft applied by a physician during surgery.

ELIGIBILITY:
Inclusion Criteria:

Torn ACL amenable to surgery

Exclusion Criteria:

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05-18 (Actual); Study Completion 2012-05-18 (Actual)

PRIMARY OUTCOMES:
Endpoints Measured at 6, 12, 18 months post op compared to pre-op

CONTACTS AND LOCATIONS:
Overall Officials: J Leith, MD, Principal Investigator — University of British Columbia